CLINICAL TRIAL: NCT06856070
Title: Evaluation of Retention and Resistance to Dislodgement of Bioflx Crowns Compared to Zirconia Crowns on Primary Molars
Brief Title: Retention of Bioflx Crowns Compared to Zirconia Crowns on Primary Molars
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, noura jamal elnoor mohamed, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RR-BFC Vs ZR
Record Dates: First submitted 2025-02-25; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Carious Primary Molars

STUDY DESIGN:
Who Masked: Participant
Masking Description: statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- (Group A: Preformed Bioflx crown) (Experimental): Kids-e-Dental LLP (ANDHERI, MUMBAI, INDIA) introduced Bioflx Crowns and claimed as the first flexible, durable, and esthetic preformed crown for primary molars. Bioflx Crowns are monochromatic, metal-free, tooth-colored crowns made up of high-strength resin polymer used in the medical device industry having high strength, flexibility, and durability. These crowns are autoclavable and are like SSC in tooth preparation as claimed by the manufacturer. Their flexibility and snap-fit technology aim to improve retention while minimizing trauma during placement
  Interventions: Other: (Group A: Preformed Bioflx crown)
- (Group B: Preformed zirconia crown) (Experimental): Zirconia crowns have been widely used in pediatric dentistry due to their high esthetic value, biocompatibility, and strength. Studies have shown that zirconia crowns exhibit superior retention due to their passive fit and resistance to fracture.
  Interventions: Other: (Group B: Preformed Zirconia crown)

INTERVENTIONS:
Other: (Group A: Preformed Bioflx crown) — prepartion:1.The mesiodistal width of the tooth will be measured using calipers and a closely fitted crown will be selected based on the measurements.
  2. The tooth will be prepared similarly to stainless steel crowns (SSCs):
  * Occlusal reduction of approximately 1-1.5 mm will be done using a diamond bur.Mesial and distal reduction of no more than 1 mm will be performed using a No. 169L diamond bur.Depending on the tooth anatomy, either no buccal and lingual reduction will be needed, or a minimal reduction will be done.
    3.All sharp line angles and corners will be smoothed to ensure proper crown fit.
    4.The crown will be checked for proper fit before cementation. It will be positioned to extend 1 mm below the gingival margin.
    5.The crown will be cemented using luting glass ionomer cement (GIC). The crown will be held with firm, constant pressure until the cement sets initially.
    6.The marginal fit will be evaluated, and necessary adjustments will be made. 7.The occlusion will be checked,
  Arms: (Group A: Preformed Bioflx crown)
Other: (Group B: Preformed Zirconia crown) — 1. Crown Selection: The mesiodistal dimension of the corresponding tooth will be measured . to select the appropriate size.2. Occlusal Reduction: The marginal ridge of adjacent teeth will be used as a reference point and a 1.5-2 mm of occlusal reduction will be performed to allow proper crown seating.3. Bucco-Lingual Reduction: The bucco-lingual wall will be reduced by approximately 1-1.5 mm using a flame-shaped diamond bur.4. Interproximal Reduction: 1 mm of interproximal reduction will be performed using a flame-shaped diamond bur such as a .368 or .330 tapered carbide bur.5. Feather Margin Preparation: Subgingival reduction of 1-2 mm will be done using a flame-shaped diamond bur, creating a feathered margin to achieve a passive fit.6. Trial Fitting of the Crown: The crown will be tried in to ensure proper adaptation. until the crown fits passively and extends sub gingivally by 1-2 mm wit.7. Glass ionomer cement will be used for cementation.
  Arms: (Group B: Preformed zirconia crown)

SUMMARY:
The goal of this clinical trial is to evaluate the retention and resistance to dislodgment of Bioflx crowns compared to zirconia crowns in the restoration of primary molars. The main question[s] it aims to answer : Is there a difference in the retention and resistance to dislodgement of BioFlx crowns compared to zirconia crowns in the restoration of primary molars?" The study will also assess the clinical performance of both types of crowns in terms of occlusal wear, gingival health, preparation time, as well as child and parental satisfaction.

DETAILED DESCRIPTION:
Primary molars play a significant role in maintaining oral function, esthetics, and space for permanent teeth, therefore, restoring decayed primary molars is a critical aspect of pediatric dentistry. Stainless steel crowns have been the standard restorative material for primary molars due to their clinical success, retention, and durability. However, the aesthetic limitations of SSCs, have been problematic, especially when patients seek more esthetically acceptable treatment options.In an attempt to address the aesthetic limitations of stainless-steel crowns, pre-veneered stainless-steel crowns were introduced featuring a thin layer of composite resin or ceramic on the outside to improve their appearance. While they provided a better aesthetic than pure stainless steel, their limitations included a tendency to wear down over time, difficulty in matching natural tooth color, and the potential for the veneer to chip or detach.Recently, zirconia crowns are preferred over pre-veneered stainless-steel crowns for their esthetic superiority, biocompatibility, and resistance to wear. They demonstrate excellent retention and durability but require significant tooth preparation, which may compromise tooth structure. Despite their advantages, zirconia crowns posed challenges such as increased cost, more complex preparation techniques, and concerns about their brittleness under certain conditions. Moreover, zirconia crowns may not be suitable for all cases, especially those involving less mineralized or structurally compromised primary molars .In 2021, Kids-e-Dental LLP introduced Bioflx Crowns and claimed as the first flexible, durable, and esthetic preformed crown for primary molars. Bioflx Crowns are monochromatic, metal-free, tooth-colored crowns made up of high-strength resin polymer used in the medical device industry having high strength, flexibility, and durability. These crowns are autoclavable and are like SSC in tooth preparation as claimed by the manufacturer. Their flexibility and snap-fit technology aim to improve retention while minimizing trauma during placement.

It is important to mention that retention is a crucial factor for the success of any dental crown. An inadequate retention can lead to crown displacement, necessitating re-treatment, and ultimately affect the long-term health of the primary tooth. While studies have demonstrated the superior esthetic properties of materials like Bioflx crowns, their clinical performance, particularly retention rates and overall longevity, require further evaluation in direct comparison to zirconia crowns .Thus, this trial aims to fill the gap in current knowledge and provide clinicians with evidence to support the choice of crown material based on retention performance, which is critical to the long-term success of pediatric restorations.

ELIGIBILITY:
Inclusion Criteria:The inclusion criteria:

1. Children aged between 4 and 8 years with primary molar that needs to be covered by crown.
2. Children who can cooperate sufficiently for the duration of the procedure, as assessed by behavior management techniques.
3. Medically healthy children (ASA I or II according to the American Society of Anesthesiologists classification).
4. Children whose parent or guardian are willing to sign an informed consent.
5. Children whose parent or guardian are willing to comply with follow-up visits. -

Exclusion Criteria:

* The exclusion criteria

  1. Molars with severe structural loss that may compromise crown retention.
  2. Children with poor oral hygiene that may contribute to higher plaque levels and affect the clinical outcomes of the crown restorations.
  3. Children with history of allergies; Known allergies to dental local anesthesia or to the materials used in Bioflx crowns.
  4. Children with any systemic conditions or disabilities that may affect their ability to participate in the study.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Retention | follow-up:T (Time): 6months interval T0: 0 T1: 3month T2: 6month
  Method of Measurement:Modified United States Public Health System criteria:Alpha: Intact Bravo:Chipped/loss of material Charlie: Complete loss of crown

SECONDARY OUTCOMES:
Occlusal wear of crown | T (Time): 6months interval T0: 0 T1: 3 month T2: 6month
  Measure by Modified United States Public Health System criteria:
  Alpha: Occlusal surface intact. Bravo: Wear of occlusal surface without tooth surface exposure Charlie: Wear of occlusal surface with
Gingival health | T (Time): 6months interval T0: 0 T1: 3month T2: 6month
  Measure by: Gingival index:
  0: healthy gum
  1. mild discoloration and edematous gingiva no bleeding on probing
  2. red oedematous and shiny gingiva bleeding on probing
  3. red oedematous and ulceration gingiva spontaneous bleeding
child and parental satisfaction | T (Time): 6months interval T0: 0T1: 3month T2: 6month
  Measure by: 5-Point likert's scale / Questionnaire:Ordinary or N/A
Preparation time | baseline
  Measure by :Stopwatch per minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.manal ahmed elshiekh Prof, Ph.D, Study Director — Cairo University
Locations (2):
- Egypt (2):
  - Faculty of Dentistry, Cairo University., Cairo, Giza Governorate
  - Faculty of Dentistry, Cairo University., Cairo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rahate I, Fulzele P, Thosar N. Comparative evaluation of clinical performance, child and parental satisfaction of Bioflx, zirconia and stainless steel crowns in pediatric patients. F1000Res. 2023 Dec 21;12:756. doi: 10.12688/f1000research.133464.2. eCollection 2023. PMID 38911945
- [Background] Patil AS, Jain M, Choubey S, Patil M, Chunawala Y. Comparative evaluation of clinical success of Stainless Steel and Bioflx crowns in primary molar - A 12 month split mouth prospective randomized clinical trial. J Indian Soc Pedod Prev Dent. 2024 Jan 1;42(1):37-45. doi: 10.4103/JISPPD.JISPPD_484_23. Epub 2024 Apr 15. PMID 38616425